CLINICAL TRIAL: NCT06187571
Title: Comparison of Conventional Therapy and Mulligan Mobilization With Movement Method in the Treatment of Shoulder Problems: A Randomized Clinical Trial
Brief Title: Mulligan Mobilization With Movement Method in the Treatment of Shoulder Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-962
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Syndrome; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWM Group (Experimental): This group received treatment with the Mulligan technique.
  Interventions: Other: CT+MWM
- CT Group (Active Comparator): This group received treatment with the conventional therapy.
  Interventions: Other: CT

INTERVENTIONS:
Other: CT+MWM — The MWM technique was applied to the MWM group in addition to the CT. The MWM technique was applied in flexion, abduction, internal rotation, and external rotation directions. The MWM technique was performed with 3 sets of 10 repetitions.
  Arms: MWM Group
Other: CT — Cold packs, electrotherapy modalities, scapular mobilization, stretching, and strengthening exercises were applied to the CT group.
  Arms: CT Group

SUMMARY:
To determine whether Mulligan mobilization with movement (MWM) and Conservative treatment CT give different results on pain, ROM, and functional activities in participants with shoulder problems.

DETAILED DESCRIPTION:
Shoulder problems are one of the common orthopedic problems. Patients with shoulder problems experience an increase in pain and a decrease in joint movement and functionality. With conventional treatment, patients' symptoms improve. However, the MWM is one of the manual therapy techniques frequently used to reduce pain in musculoskeletal system problems. It is extremely important to evaluate patients' functionality after rehabilitation. Although there are studies comparing the effect of MWM in the literature, studies evaluating patient-specific functionality are also limited.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Having any shoulder problems (impingement, rotator cuff syndrome, glenohumeral joint problems, etc.),
* Having a history of shoulder pain lasting at least 3 months, and volunteering to participate in the study.

Exclusion Criteria:

* Having systemic or degenerative disease, a neurological disease, and
* Having more than one upper extremity pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Shoulder pain | through study completion, an average of 6 month
  The Numeric Pain Rating Scale was used to evaluate shoulder pain. The patient was asked to mark the point corresponding to the pain between 0 and 10. The higher the score, the higher the pain.

SECONDARY OUTCOMES:
ROM | through study completion, an average of 6 month
  Shoulder flexion, abduction, internal and external rotation were measured using a Universal goniometer.As the angle increases, the joint range of motion increases.
Patient Specific Functional Scale | through study completion, an average of 6 month
  In the patient-specific activity scale, depending on the current pathology, the physiotherapist asks the patient three or five activities that he or she finds difficult to do. The patient is asked to score the activity between 0-10 points. The total score is determined by averaging the activity scores, with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)